CLINICAL TRIAL: NCT04894812
Title: The Effect of Vestibular Stimulation Along With Neurodevelopmental Technique on Motor Functions of Children With Hemiplegic Cerebral Palsy
Brief Title: Vestibular and Motor Functions in Children With Hemiplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/00757 Anam Tariq
Record Dates: First submitted 2021-05-19; First posted 2021-05-20 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Cerebral Palsy; Hemiplegic Cerebral Palsy
Keywords: motor activity; spasticity; vestibular stimulation
MeSH Terms: conditions — Cerebral Palsy; Motor Activity; Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Neurodevelopmental Treatment. Total duration of treatment will be 20 minutes, 3 sessions per for 3 months
  Interventions: Other: Neurodevelopmental technique
- Group B (Experimental): Neurodevelopmental Technique and Vestibular stimulation. Total duration of treatment will be 50 minutes (20 min NDT+ 30 MIN VS) 3 sessions per week for 3 months.
  Interventions: Other: Neurodevelopmental technique

INTERVENTIONS:
Other: Neurodevelopmental technique — 1. st month: postural maintenance; exercises with weight on forearms and hands, in sitting, crawling, semi-kneeling and standing positions with support from therapist.
  2. nd month: balance and corrective reactions; using CP ball and tilt board.
  3. rd month: ambulation training; appropriate to motor development level (crawling, creeping, walking in a semi-kneeling position and walking between parallel bars).

SUMMARY:
As many researches have been conducted to see the effects of vestibular system activation on gross motor activities of children with cerebral palsy but there are limited researches on improvement of motor abilities of hemiplegic cerebral palsy child using UEU or BOSU ball or treadmill in a single study. There is lack of research on vestibular stimulation in hemiplegic cerebral palsy along with neurodevelopmental treatment.

This study will improve the gross motor activities of children with hemiplegic cerebral palsy. It will broaden up the ways for physical therapist to deal with this type of cerebral palsy (hemiplegic).

DETAILED DESCRIPTION:
There are various therapeutic approaches that are used to improve motor activities and postural control in CP child. Among these approaches vestibular stimulation is used to improve neuromotor development by different sensory stimulation techniques. It has shown positive effects on motor control of CP child. It also influences all sensory experiences and is an exercise based approach.

ELIGIBILITY:
Inclusion Criteria:

* Age: 3 years to 12 years
* Gender: Both Male and female
* Children with Spastic Hemiplegic CP scoring 1,1+ and 2 on Modified Ashworth scale
* Level III and IV on GMFCS (Gross Motor Function Classification System)

Exclusion Criteria:

* Children with other types of Cerebral Palsy (diplegia, quadriplegia etc)
* Children with other Abnormalities and pathologies (delayed milestones, hydrocephalous, epilepsy etc)
* Children Undergone any kind of surgery (cardiac, shunt placement, orthopedic etc)
* Children with any other neurological deficits (spina bifida etc)
* Children with conditions in which vestibular stimulation is not allowed (paroxysmal positional vertigo or vestibular neuritis, Meniere's disease, migraine-associated vertigo, and childhood vertigo).

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
GMFM-88 | 12 weeks
  It is a Standardized Observational Instrument designed and validated to measure change in gross motor function over time in children with Cerebral Palsy. The GMFM-88 item scores can be summed to calculate raw and percent scores for each of the five GMFM dimensions of interest, selected goal areas and a total GMFM-88 score.

SECONDARY OUTCOMES:
Modified Ashworth Scale | 12 weeks
  The purpose of the Modified Ashworth Scale is to measure spasticity in patients who have lesions of the CNS or neurological disorders. The MAS is a quick and easy measure that can assist a clinician's assessment of spasticity during passive soft-tissue stretching.

CONTACTS AND LOCATIONS:
Overall Officials: Mirza Obaid Baig, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Institute of Pediatric Habilitation and Rehabilitation IPH, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tramontano M, Medici A, Iosa M, Chiariotti A, Fusillo G, Manzari L, Morelli D. The Effect of Vestibular Stimulation on Motor Functions of Children With Cerebral Palsy. Motor Control. 2017 Jul;21(3):299-311. doi: 10.1123/mc.2015-0089. Epub 2016 Aug 19. PMID 27633076
- [Background] Bangash AS, Hanafi MZ, Idrees R, Zehra N. Risk factors and types of cerebral palsy. J Pak Med Assoc. 2014 Jan;64(1):103-7. PMID 24605730
- [Background] Labaf S, Shamsoddini A, Hollisaz MT, Sobhani V, Shakibaee A. Effects of Neurodevelopmental Therapy on Gross Motor Function in Children with Cerebral Palsy. Iran J Child Neurol. 2015 Spring;9(2):36-41. PMID 26221161